CLINICAL TRIAL: NCT03941405
Title: Albumin for Management of Hypervolemic Hyponatremia in Patients With Decompensated Cirrhosis. A Proof of Concept Study.
Brief Title: Albumin for Management of Hypervolemic Hyponatremia (AlbuCAT)
Acronym: AlbuCAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-000302-29
Record Dates: First submitted 2019-03-28; First posted 2019-05-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hyponatremia With Excess Extracellular Fluid Volume; Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Albumins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No treatment (No Intervention): No treatment.
- Albumin treatment (Experimental): one dose per day of a 40g albumin g/l gram(s)/litre for 10 days.
  Interventions: Drug: Albumin treatment

INTERVENTIONS:
Drug: Albumin treatment — one dose per day of a 40g albumin g/l gram(s)/litre for 10 days. resolution of hyponatremia, defined as an increase in serum sodium of more than 5 mEq/L with a final value > 130 mEq/L, maintained for at least 48 consecutive hours during the 10-day treatment period
  Other Names: Human Albumin Grifols 200 g/l, solution for infusion
  Arms: Albumin treatment

SUMMARY:
resolution of hyponatremia, defined as an increase in serum sodium of more than 5 mEq/L with a final value > 130 mEq/L, maintained for at least 48 consecutive hours during the 10-day treatment period

ELIGIBILITY:
Inclusion Criteria:

* Patients included into the study must meet all the following criteria:

This study will include patients with liver cirrhosis and hypervolemic hyponatremia (serum sodium<130 mEq/L) admitted to hospital for any decompensation of the disease. Patients will be enrolled if hyponatremia persists after 3 days of diuretic withdrawal and fluid restriction. Women of child-bearing potential must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods, including intrauterine device, bilateral tubal occlusion or a vasectomized partner. Hormonal contraceptive methods will be avoided due to the risk of adverse events and impairment of liver function.

Exclusion Criteria:

1. Patients with Acute kidney injury 1B or higher;
2. Chronic kidney disease grade 3a or higher, defined as glomerular filtration rate <60ml/min for three months and markers of kidney damage (one or more): Albuminuria (Albumin excretion rate > 30 mg/24h; Albumin-to-creatinine ratio > 30 mg/g), Urine sediment abnormalities, Electrolyte and other abnormalities due to tubular disorders, Electrolyte and other abnormalities due to tubular disorders, Abnormalities detected by histology or Structural abnormalities detected by imaging.
3. Previous kidney or liver transplant;
4. Active infection apart from spontaneous bacterial peritonytis based on positive culture (blood, urine, sputum or other samples) or by the following criteria:

   1. Urinary infections: signs of systemic inflammation and more than 10 leukocytes per high-power field in urine;
   2. Pneumonia: compatible symptoms (cough, purulent sputum, chest pain, shortness of breath) and presence of new infiltrates on chest x-ray;
   3. Skin/soft tissue infection: physical exam findings of swelling, erythema, heat and tenderness in the skin;
   4. Acute cholangitis: signs of systemic inflammation1, compatible symptoms (right upper quadrant pain and jaundice) and radiological data of biliary obstruction, analytical data of cholestasis;
   5. Suspected bacterial infection: signs of systemic inflammation1 but no identifiable origin of this infection (polymorphonuclear cells in ascitic and pleural fluid < 250/mm3, normal urine sediment and chest Xray) After 48 hours of appropriate antibiotic treatment patients can be enrolled.
5. Spontaneous bacterial peritonitis.
6. Hypo or hyperthyroidism not controlled under adequate treatment.
7. Associated heart failure, defined as a New York Heart Association (NYHA) classification III or IV or heart failure with reduced ejection fraction (LVEF<40%). Previously known structural cardiomyopathy including ischemic cardiomyopathy, restrictive cardiomyopathy or valvular cardiomyopathy.
8. Hepatocellular carcinoma beyond Milan criteria.
9. Severe alcoholic hepatitis defined by Maddrey score ≥32 and/or MELD score ≥ 20
10. ACLF with two or more organ failures
11. Treatment with diuretics (furosemide or spironolactone), albumin infusion, somatostatin or terlipresin in the previous 3 days.
12. Symptomatic hyponatremia (manifested by cardio-respiratory distress, abnormal and deep somnolence, seizures or coma) with serum sodium below 120 mEq/L.
13. Previous known hypersensitivity to human albumin
14. Refuse to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Resolution of hyponatremia | for at least 48 consecutive hours during the 10-day treatment
  defined as an increase in serum sodium of more than 5 mEq/L with a final value > 130 mEq/L

SECONDARY OUTCOMES:
partial resolution of hyponatremia | maintained for at least 48 consecutive hours during the 10-day treatment period.
  defined as an increase in serum sodium of more than 5meq/L with a final value below 130meq/L,
Evaluation of systemic hemodynamics | levels at day 0, at day 5 and at day 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days) of the study period.
  mean arterial pressure
kidney function | levels at day 0, 5 and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  measurement of creatinine levels
Effects on the inflammatory profile | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  evaluation of PCR of plasma cytokines by using a multiplex kit including plasmatic cytokines related to immune response. This multiplex test will be performed at day 0 and day 10 of the study period (or at the end of study in case of early termination).
Effects on neurocognitive function and quality | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  PHES questionnaire
Effects on brain water content | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  performance of aMagnetic Resonance Spectroscopy (MRS)
Effects of albumin administration on liver phagocytic capacity | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  Effects of albumin administration on liver phagocytic capacity as assessed by performance of hepatic SPECT with 99mTc-phytate at day 0 and 10 (or at the end of study in case of early termination).
Effects on phagocytic capacity and inflammatory response of peripheral monocytes | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  Effects on phagocytic capacity and inflammatory response of peripheral monocytes will be assessed by performance specific tests (Phagotest and Phagoburst) evaluating the in vitro phagocytic capacity and burst response. Monocytes will be isolated and analysed at day 0 and at day 10 of the study period (or at the end of study in case of early termination).
Effects of albumin administration of microbiome composition | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  Effects of albumin administration of microbiome composition as assessed by analysis of microbiome composition at day 0 and 10 of the study period (or at the end of study in case of early termination).
Effects of albumin administration on development of infections, development of complications of cirrhosis and survival. | levels at day 0, and 10 (or at the end of study in case of early termination due to primary endpoint reach from day 0 up to 10 days).
  Effects of albumin administration on development of infections, development of complications of cirrhosis and survival.
Effects of albumin administration on serum albumin levels | levels at day 0, 5, 10, 28 and 90 of study period.
  Effects of albumin administration on serum albumin levels assessed by measurement of mEq/L serum albumin levels at day 0, 5, 10, 28 and 90 of study period.
evaluate treatment-related serious adverse events | visit day 1,2,3,4,5,6,7,8,9,28 and 90
  To evaluate treatment-related serious adverse events during the treatment period

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital Moises Broggi, Barcelona, Catalonia
  - Hospital Parc Taulí, Sabadell, Catalonia